CLINICAL TRIAL: NCT03484702
Title: A Phase 2, Single-arm, Multi-center Trial to Determine the Efficacy and Safety of JCAR017 in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma or With Other Aggressive B-Cell Malignancies
Brief Title: Trial to Determine the Efficacy and Safety of JCAR017 in Adult Participants With Aggressive B-Cell Non-Hodgkin Lymphoma
Acronym: TRANSCENDWORLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCAR017-BCM-001; U1111-1209-4055 (Other Grant/Funding Number: WHO); 2017-000106-38 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkin lymphoma; Aggressive B-cell non-Hodgkin lymphoma; Diffuse large B-cell lymphoma; Relapse / refractory lymphoma; Transplant not eligible; High-grade B-cell lymphoma; Primary central nervous system lymphoma; Transformed follicular lymphoma; Follicular lymphoma Grade 3B; JCAR017; Liso-Cel
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Administration of JCAR017 (Experimental)
  Interventions: Drug: JCAR017

INTERVENTIONS:
Drug: JCAR017 — Specified dose on specified days
  Other Names: Lisocabtagene Maraleucel (liso-cel)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of JCAR017 in participants with aggressive B-cell non-Hodgkin lymphoma (B-NHL)

DETAILED DESCRIPTION:
This is a study to determine the efficacy and safety of JCAR017 in adult participants with aggressive B-cell NHL. The study will enroll participants in Europe and Japan with diffuse large B-cell lymphoma (DLBCL) not otherwise specified (NOS; de novo or transformed follicular lymphoma [tFL]), high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (HGBL), follicular lymphoma Grade 3B (FL3B), and primary central nervous system lymphoma (PCNSL). Participants with secondary central nervous system (CNS) involvement are allowed.

Once enrolled, participants will undergo leukapheresis to enable JCAR017 cell product generation. Upon successful JCAR017 cell product generation, participants will receive lymphodepleting chemotherapy followed by infusion of JCAR017. JCAR017 will be administered by intravenous infusion. Participants will be followed for approximately 2 years after their JCAR017 infusion for safety, disease status, survival and health-related quality of life.

Delayed adverse events following exposure to gene modified T cells will be assessed and long-term persistence of these modified T cells will continue to be monitored under a separate long-term follow-up protocol for up to 15 years after JCAR017 infusion as per competent authority guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of diagnosis at last relapse
* Adequate organ function
* Adequate vascular access for leukapheresis procedure

Exclusion Criteria:

* Prior history of malignancies, other than aggressive relapsed/refractory Non-Hodgkin Lymphoma, unless the participant has been in remission for ≥ 2 years with the exception of non-invasive malignancies
* Received previous CD19-targeted therapy
* Progressive vascular tumor invasion, thrombosis, or embolism

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- Local Institution - 101, Vienna, Austria
- Local Institution - 351, Ghent, Belgium
- Local Institution - 551, Helsinki, Finland
- France (3):
  - Local Institution - 202, Lille
  - Local Institution - 203, Paris
  - Local Institution - 201, Pierre-Bénite
- Germany (5):
  - Local Institution - 151, Cologne
  - Local Institution - 152, Dresden
  - Local Institution - 155, Heidelberg
  - Local Institution - 154, München
  - Local Institution - 153, Ulm
- Italy (2):
  - Local Institution - 402, Milan
  - Local Institution - 401, Torino
- Japan (2):
  - Local Institution - 601, Chuo-ku, Tokyo
  - Local Institution - 602, Minato-ku, Tokyo
- Local Institution - 301, Rotterdam, Netherlands
- Local Institution - 451, Barcelona, Spain
- Local Institution - 251, Bern, Switzerland
- United Kingdom (2):
  - Local Institution - 502, Manchester, Lancashire
  - Local Institution - 501, London

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the pretreatment period participants underwent leukapheresis to enable JCAR017 cell product generation. Upon successful JCAR017 cell product generation, participants entered the treatment period and received lymphodepleting chemotherapy followed by infusion of JCAR017.
  Cohort 6 was planned but subsequently removed from the study. No participants were enrolled into Cohort 6.
Groups:
- Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy; Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy; Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2; Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma; Cohort 5: Primary Central Nervous System Lymphoma; Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting: JCAR017 was infused at a dose of 100 x 10^6 JCAR017-positive transfected viable T cells (50 × 10^6 CD8+ CAR+ T cells and 50 × 10^6 CD4+ CAR+ T cells), on Day 1 (2 to 7 days after completion of Lymphodepleting chemotherapy).
Period: Pre-Treatment Period - Leukapheresis
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Started (Underwent Leukapheresis) | 45 | 32 | 14 | 4 | 7 | 11
Completed | 43 | 27 | 12 | 1 | 5 | 10
Not Completed | 2 | 5 | 2 | 3 | 2 | 1
Period: Treatment Period
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Started (Started lymphodepleting chemotherapy.) | 43 | 27 | 12 | 1 | 5 | 10
JCAR017 Treated Set (Received conforming JCAR017 cell product.) | 36 | 27 | 10 | 1 | 5 | 9
Completed | 39 | 24 | 12 | 1 | 5 | 9
Not Completed | 4 | 3 | 0 | 0 | 0 | 1
Not completed — Death | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Withdrew from Study | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting | Total
Number analyzed (Participants) | 45 | 32 | 14 | 4 | 7 | 11 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (10.60) | 73.3 (5.50) | 57.6 (10.08) | 63.5 (21.11) | 57.0 (5.74) | 58.1 (12.47) | 63.3 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 6 | 1 | 3 | 4 | 42
  Male | 30 | 19 | 8 | 3 | 4 | 7 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 0 | 1 | 0 | 1 | 10
  Not Hispanic or Latino | 29 | 22 | 14 | 2 | 5 | 7 | 79
  Unknown or Not Reported | 9 | 9 | 0 | 1 | 2 | 3 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 14 | 0 | 0 | 0 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 37 | 19 | 0 | 3 | 5 | 7 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 0 | 1 | 2 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per Independent Review Committee in Cohorts 1, 2 and 3
Description: Overall response rate (ORR) by Independent Review Committee (Cohorts 1, 2, 3). ORR is the percent of participants with best overall response of complete response (CR) or partial response (PR).
  Complete response via PET-CT:
  * Lymph nodes/extralymphatic: Score 1, 2, 3a with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease
  Complete response via CT scan:
  * Lymph nodes/extralymphatic: Target nodes/nodal masses ≤ 1.5 cm longest transverse diameter.
  * Nonmeasured lesion: No
  * New lesions: No
  * Bone marrow: Normal
  Partial response via PET-CT:
  * Lymph nodes/extralymphatic: Score 4, 5b, reduced uptake from baseline
  * New lesions: No
  * Bone marrow: Residual uptake higher than normal, reduced from baseline
  Partial response via CT scan:
  * Lymph nodes/extralymphatic: 50% decrease in sum of diameters of <= 6 target measurable nodes/extranodal sites
  * Nonmeasured lesion: No
  * Organ enlargement: Spleen length decreased > 50%
  * New lesions: No
Time Frame: From JCAR017 infusion until disease progression, end of study, the start of another anticancer therapy, or hemopoietic stem cell transplant (HSCT) (up to approximately 63 months)
Population: All participants in the JCAR017 treated set. Prespecified to be reported for cohorts 1,2, and 3 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2
Number analyzed (Participants) | 36 | 27 | 10
Percent of Participants | 61.1 [43.5 to 76.9] | 63.0 [42.4 to 80.6] | 70.0 [34.8 to 93.3]

2. Primary Outcome: Overall Response Rate (ORR) Per Investigator in Cohort 4
Description: Overall response rate (ORR) is the percent of participants with best overall response of complete response (CR) or partial response (PR).
  Complete response via PET-CT:
  * Lymph nodes/extralymphatic: Score 1, 2, 3a with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease
  Complete response via CT scan:
  * Lymph nodes/extralymphatic: Target nodes/nodal masses ≤ 1.5 cm longest transverse diameter.
  * Nonmeasured lesion: None
  * New lesions: No
  * Bone marrow: Normal
  Partial response via PET-CT:
  * Lymph nodes/extralymphatic: Score 4, 5b, reduced uptake from baseline
  * New lesions: None
  * Bone marrow: Residual uptake higher than normal, reduced from baseline
  Partial response via CT scan:
  * Lymph nodes/extralymphatic: 50% decrease in sum of diameters of <= 6 target measurable nodes/extranodal sites
  * Nonmeasured lesion: None/normal
  * Organ enlargement: Spleen length decreased > 50%
  * New lesions: No
Time Frame: as for outcome 1
Population: All participants in the JCAR017 treated set. Prespecified to be reported for cohort 4 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma
Number analyzed (Participants) | 1
Percent of Participants | 100 [100 to 100]

3. Primary Outcome: Overall Response Rate (ORR) Per Investigator in Cohort 5
Description: Overall response rate (ORR) determined by Investigator assessment after JCAR017 infusion. The ORR is the percent of participants with best overall response (BOR) of either complete response (CR), complete response unconfirmed (Cru) or partial response (PR).
  Complete response (CR):
  * Brain imaging: No contrast enhancement
  * Corticosteroid dose: None
  * Eye examination: Normal
  * Cerebrospinal fluid cytology: Negative
  Complete response unconfirmed (CRu):
  * Brain imaging: No contrast enhancement, Minimal abnormality
  * Corticosteroid dose: Any
  * Eye examination: Normal, minor RPE abnormality
  * Cerebrospinal fluid cytology: Negative
  Partial response (PR):
  * Brain imaging: 50% decrease in enhancing tumor, no contrast enhancement.
  * Corticosteroid dose: Irrelevant
  * Eye examination: Minor RPE abnormality, decrease in vitreous cells or retinal infiltrate.
  * Cerebrospinal fluid cytology: Negative, persistent or suspicious
Time Frame: as for outcome 1
Population: All participants in the JCAR017 treated set. Prespecified to be reported for cohort 5 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 5: Primary Central Nervous System Lymphoma
Number analyzed (Participants) | 5
Percent of Participants | 80.0 [28.4 to 99.5]

4. Primary Outcome: Number of Participants With Adverse Events in Cohort 7
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE. Graded according to NCI CTCAE (Version 4.03) guidelines where grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life threatening, grade 5 = death.
Time Frame: From leukapheresis to end of study (up to approximately 63 months)
Population: All participants in the JCAR017 treated set. Prespecified to be reported for cohort 7 only
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 9
Participants
  AEs occurring between leukapheresis and lymphodepleting chemotherapy (LDC) | 0
  AEs occurring between LDC and JCAR017 infusion | 2
  AEs occurring between JCAR017 infusion and Day 30 | 9
  AEs occurring between Day 31 and Day 90 | 7
  AEs occurring between Day 91 and end of study | 7

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) in Cohort 7
Description: A serious adverse event (SAE) is defined as any adverse event (AE) occurring at any dose that:
  * Results in death;
  * Is life-threatening (ie, in the opinion of the Investigator, the participant is at immediate risk of death from the AE);
  * Requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay).
  * Results in persistent or significant disability/incapacity (a substantial disruption of the participant's ability to conduct normal life functions);
  * Is a congenital anomaly/birth defect;
  * Constitutes an important medical event. Graded according to NCI CTCAE (Version 4.03) guidelines where grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life threatening, grade 5 = death.
Time Frame: From leukapheresis to end of study (up to approximately 63 months)
Population: All participants in the JCAR017 treated set. Prespecified to be reported for cohort 7 only
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 9
Participants
  SAEs occurring between leukapheresis and lymphodepleting chemotherapy (LDC) | 0
  SAEs occurring between LDC and JCAR017 infusion | 0
  SAEs occurring between JCAR017 infusion and Day 30 | 1
  SAEs occurring between Day 31 and Day 90 | 0
  SAEs occurring between Day 91 and end of study | 1

6. Primary Outcome: Number of Participants With Increase From Baseline in Select Hematology Parameters - Cohort 7
Description: JCAR017 treatment-emergent laboratory abnormalities are defined as an abnormality that, compared to baseline, worsens by at least one grade after JCAR017 infusion. The baseline value is defined as the last available recorded value on or prior to the date of JCAR017 infusion. Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Life-threatening), Grade 5 (Death).
Time Frame: At Baseline and Day 29 after JCAR017 infusion
Population: All participants in the JCAR017 treated set with available baseline and Day 29 hematology results. Prespecified to be reported for cohort 7 only
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 9
Participants
  Leukocytes (10^9/L) - Day 29 | 0
  Neutrophils, Segmented (10^9/L) - Day 29: number analyzed (Participants) | 8
  Neutrophils, Segmented (10^9/L) - Day 29 | 2
  Platelets (10^9/L) - Day 29 | 5
  Activated Partial Thromboplastin Time (sec) - Day 29 | 0
  Prothrombin Intl. Normalized Ratio - Day 29 | 1

7. Primary Outcome: Number of Participants With Increase From Baseline in Select Serum Chemistry Parameters - Cohort 7
Description: as for outcome 6
Time Frame: At Baseline and Day 29 after JCAR017 infusion
Population: All participants in the JCAR017 treated set with available baseline and Day 29 serum chemistry results. Prespecified to be reported for cohort 7 only
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 9
Participants
  Albumin (g/L) - Day 29 | 0
  Phosphate (mmol/L) - Day 29: number analyzed (Participants) | 8
  Phosphate (mmol/L) - Day 29 | 0
  Alkaline Phosphatase (U/L) - Day 29 | 0
  Alanine Aminotransferase (U/L) - Day 29 | 0
  Aspartate Aminotransferase (U/L) - Day 29 | 1
  Bilirubin (umol/L) - Day 29 | 0
  Creatinine (umol/L) - Day 29 | 7
  Triglycerides (mmol/L) - Day 29 | 3
  Urate (umol/L) - Day 29 | 0

8. Secondary Outcome: Number of Participants With Adverse Events in Cohorts 1, 2, 3, 4, and 5
Description: as for outcome 4
Time Frame: From leukapheresis to end of study (up to approximately 63 months)
Population: All participants in the JCAR017 treated set. Prespecified to be reported for Cohorts 1, 2, 3, 4, and 5 only
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma
Number analyzed (Participants) | 36 | 27 | 10 | 1 | 5
Participants
  AEs occurring between leukapheresis and lymphodepleting chemotherapy (LDC) | 5 | 5 | 0 | 0 | 0
  AEs occurring between LDC and JCAR017 infusion | 29 | 23 | 8 | 0 | 4
  AEs occurring between JCAR017 infusion and Day 30 | 36 | 26 | 10 | 1 | 5
  AEs occurring between Day 31 and Day 90: number analyzed (Participants) | 35 | 27 | 10 | 1 | 5
  AEs occurring between Day 31 and Day 90 | 25 | 10 | 8 | 1 | 3
  AEs occurring between Day 91 and end of study: number analyzed (Participants) | 32 | 23 | 8 | 1 | 5
  AEs occurring between Day 91 and end of study | 10 | 9 | 7 | 0 | 2

9. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) in Cohorts 1, 2, 3, 4, and 5
Description: A serious adverse event (SAE) is defined as any adverse event (AE) occurring at any dose that:
  * Results in death;
  * Is life-threatening (ie, in the opinion of the Investigator, the participant is at immediate risk of death from the AE);
  * Requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay).
  * Results in persistent or significant disability/incapacity (a substantial disruption of the participant's ability to conduct normal life functions);
  * Is a congenital anomaly/birth defect;
  * Constitutes an important medical event. Graded according to NCI CTCAE (Version 4) guidelines where grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life threatening, grade 5 = death.
Time Frame: From leukapheresis to end of study (up to approximately 63 months)
Population: All participants in the JCAR017 treated set. Prespecified to be reported for cohorts 1, 2, 3, 4, and 5 only
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma
Number analyzed (Participants) | 36 | 27 | 10 | 1 | 5
Participants
  SAEs occurring between leukapheresis and lymphodepleting chemotherapy (LDC) | 0 | 1 | 0 | 0 | 0
  SAEs occurring between LDC and JCAR017 infusion | 1 | 0 | 0 | 0 | 0
  SAEs occurring between JCAR017 infusion and Day 30 | 16 | 7 | 0 | 0 | 1
  SAEs occurring between Day 31 and Day 90: number analyzed (Participants) | 35 | 27 | 10 | 1 | 5
  SAEs occurring between Day 31 and Day 90 | 7 | 3 | 2 | 0 | 1
  SAEs occurring between Day 91 and end of study: number analyzed (Participants) | 32 | 23 | 8 | 1 | 5
  SAEs occurring between Day 91 and end of study | 5 | 3 | 1 | 0 | 0

10. Secondary Outcome: Number of Participants With Increase From Baseline in Select Hematology Parameters - Cohorts 1, 2, 3, 4, and 5
Description: JCAR017 treatment-emergent laboratory abnormalities are defined as an abnormality that, compared to baseline, worsens by at least one grade after JCAR017 infusion. The baseline value is defined as the last available recorded value on or prior to the date of JCAR017 infusion. Grade 1 = Mild, Grade 2 =Moderate, Grade 3 =Severe, Grade 4 =Life-threatening, Grade 5 =Death.
Time Frame: At Baseline and Day 29 after JCAR017 infusion
Population: All participants in the JCAR017 treated set with available baseline and Day 29 hematology results. Prespecified to be reported for cohorts 1, 2, 3, 4, and 5 only
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma
Number analyzed (Participants) | 33 | 21 | 10 | 1 | 5
Participants
  Leukocytes (10^9/L) - Day 29 | 4 | 2 | 1 | 0 | 1
  Neutrophils, Segmented (10^9/L) - Day 29 | 11 | 6 | 3 | 0 | 1
  Platelets (10^9/L) - Day 29: number analyzed (Participants) | 29 | 20 | 10 | 1 | 5
  Platelets (10^9/L) - Day 29 | 13 | 8 | 9 | 1 | 3
  Activated Partial Thromboplastin Time (sec) - Day 29: number analyzed (Participants) | 32 | 18 | 8 | 1 | 3
  Activated Partial Thromboplastin Time (sec) - Day 29 | 0 | 1 | 1 | 0 | 1
  Prothrombin Intl. Normalized Ratio - Day 29: number analyzed (Participants) | 32 | 21 | 8 | 1 | 3
  Prothrombin Intl. Normalized Ratio - Day 29 | 1 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Increase From Baseline in Select Serum Chemistry Parameters - Cohorts 1, 2, 3, 4, and 5
Description: as for outcome 10
Time Frame: At Baseline and Day 29 after JCAR017 infusion
Population: All participants in the JCAR017 treated set with available baseline and Day 29 serum chemistry results. Prespecified to be reported for cohorts 1, 2, 3, 4, and 5 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma
Number analyzed (Participants) | 35 | 24 | 10 | 1 | 4
Participants
  Albumin (g/L) - Day 29 | 0 | 0 | 0 | 0 | 0
  Phosphate (mmol/L) - Day 29 | 0 | 1 | 0 | 0 | 0
  Alkaline Phosphatase (U/L) - Day 29 | 2 | 1 | 0 | 0 | 1
  Alanine Aminotransferase (U/L) - Day 29 | 10 | 3 | 1 | 0 | 2
  Aspartate Aminotransferase (U/L) - Day 29: number analyzed (Participants) | 35 | 23 | 10 | 1 | 4
  Aspartate Aminotransferase (U/L) - Day 29 | 6 | 3 | 1 | 0 | 3
  Bilirubin (umol/L) - Day 29: number analyzed (Participants) | 34 | 23 | 10 | 1 | 4
  Bilirubin (umol/L) - Day 29 | 2 | 0 | 0 | 0 | 0
  Creatinine (umol/L) - Day 29 | 23 | 20 | 6 | 1 | 3
  Triglycerides (mmol/L) - Day 29 | 10 | 6 | 2 | 0 | 2
  Urate (umol/L) - Day 29 | 1 | 0 | 0 | 0 | 0

12. Secondary Outcome: Overall Response Rate (ORR) in Cohort 7
Description: ORR by Independent Review Committee. ORR is the percent of participants with best overall response of complete response (CR) or partial response (PR).
  Complete response via PET-CT:
  * Lymph nodes/extralymphatic: Score 1, 2, 3a with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease
  Complete response via CT scan:
  * Lymph nodes/extralymphatic: Target nodes/nodal masses ≤ 1.5 cm longest transverse diameter.
  * Nonmeasured lesion: None
  * New lesions: No
  * Bone marrow: Normal
  Partial response via PET-CT:
  * Lymph nodes/extralymphatic: Score 4, 5b, reduced uptake from baseline
  * New lesions: None
  * Bone marrow: Residual uptake higher than normal, reduced from baseline
  Partial response via CT scan:
  * Lymph nodes/extralymphatic: 50% decrease in sum of diameters of <= 6 target measurable nodes/extranodal sites
  * Nonmeasured lesion: None/normal
  * Organ enlargement: Spleen length decreased > 50%
  * New lesions: No
Time Frame: as for outcome 1
Population: All participants in the JCAR017 treated set. Prespecified to be reported for cohort 7 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 9
Percent of Participants | 88.9 [51.8 to 99.7]

13. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete response rate is defined as percentage of participants achieving a best overall response of complete response.
  Complete response via PET-CT:
  * Lymph nodes/extralymphatic: Score 1, 2, 3a with/without residual mass on 5-point scale
  * New lesions: No
  * Bone marrow: No FDG-avid disease
  Complete response via CT scan:
  * Lymph nodes/extralymphatic: Target nodes/nodal masses ≤ 1.5 cm longest transverse diameter.
  * Nonmeasured lesion: None
  * New lesions: No
  * Bone marrow: Normal
  Complete response (CR) (Cohort 5):
  * Brain imaging: No contrast enhancement
  * Corticosteroid dose: None
  * Eye examination: Normal
  * Cerebrospinal fluid cytology: Negative
  Complete response unconfirmed (CRu) (Cohort 5):
  * Brain imaging: No contrast enhancement, Minimal abnormality
  * Corticosteroid dose: Any
  * Eye examination: Normal, minor RPE abnormality
  * Cerebrospinal fluid cytology: Negative
Time Frame: as for outcome 1
Population: All participants in the JCAR017 treated set.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 36 | 27 | 10 | 1 | 5 | 9
Percent of Participants | 33.3 [18.6 to 51.0] | 48.1 [28.7 to 68.1] | 50.0 [18.7 to 81.3] | 0 [0 to 0] | 0 [0 to 0] | 88.9 [51.8 to 99.7]

14. Secondary Outcome: Event Free Survival (EFS)
Description: Event-free survival is from JCAR017 infusion to death from any cause, progressive disease, or starting a new anticancer therapy. If a participant did not have an EFS event prior to data cutoff, EFS was censored at last disease assessment.
  Progressive disease (PD):
  * Target nodes/nodal masses: PPD progression.
  * Extranodal lesion: LDi > 1.5 cm and increase by ≥ 50% from PPD nadir.
  * Splenomegaly: > 50% of prior increase from baseline or by at least 2 cm from baseline.
  * Nonmeasured lesions: New or clear progression.
  * New lesions: Regrowth of previously resolved lesions.
  * Bone marrow: New or recurrent
  Progressive Disease (Cohort 5):
  * Brain imaging: > 25% increase in enhancing lesion from baseline or best response.
  * Eye Exam: Increased vitreous cell counts or progressive retinal or optic nerve infiltration.
  * New lesion or site of disease
Time Frame: From JCAR017 infusion to death due to any reason, progressive disease, or starting a new anticancer therapy (up to approximately 63 months).
Population: All participants in the JCAR017 treated set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 36 | 27 | 10 | 1 | 5 | 9
Months | 2.99 [2.60 to 5.22] | 3.12 [1.97 to 7.36] | 6.33 [0.56 to NA] — Insufficient number of events to calculate upper limit of the CI using the K-M method. | 23.95 [23.95 to 23.95] | 14.23 [0.76 to 24.02] | NA [5.65 to NA] — Insufficient number of events to calculate median and upper limit of the CI using the K-M method.

15. Secondary Outcome: Progression Free Survival (PFS) Using European Medicines Agency (EMA) Criteria
Description: Progression-free survival is defined as the interval from the date of JCAR017 infusion to progressive disease or death due to any cause, whichever occurred first. Per European Medicines Agency (EMA) criteria, participants who did not experience progressive disease and who did not die before the data cutoff date were censored at the time of the last visit with adequate response assessment when the participants were known not to have progressed.
  Estimated using Kaplan-Meier product-limit estimates.
Time Frame: From JCAR017 infusion to progressive disease or death due to any reason, whichever occurred first (up to approximately 63 months)
Population: All participants in the JCAR017 treated set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 36 | 27 | 10 | 1 | 5 | 9
Months | 2.99 [2.76 to 5.22] | 3.12 [1.97 to 7.36] | 6.33 [0.56 to NA] — Insufficient number of events to calculate upper limit of the CI using the K-M method. | 14.23 [0.76 to 24.02] | 23.95 [23.95 to 23.95] | NA [5.65 to NA] — Insufficient number of events to calculate median and upper limit of the CI using the K-M method.

16. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the interval from the date of JCAR017 infusion to the date of death due to any reason. Data from surviving participants was censored at the last time that the participant was known to be alive.
  Estimated using Kaplan-Meier product-limit estimates.
Time Frame: From the date of JCAR017 infusion to the date of death due to any reason (up to approximately 63 months).
Population: All participants in the JCAR017 treated set.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 36 | 27 | 10 | 1 | 5 | 9
Months | 15.84 [5.82 to 23.95] | 16.82 [4.27 to NA] — Insufficient number of events to calculate upper limit of the CI using the K-M method. | 14.72 [1.71 to NA] — Insufficient number of events to calculate upper limit of the CI using the K-M method. | 31.74 [31.74 to 31.74] | 14.23 [4.30 to NA] — Insufficient number of events to calculate upper limit of the CI using the K-M method. | NA [11.60 to NA] — Insufficient number of events to calculate median and upper limit of the CI using the K-M method.

17. Secondary Outcome: Duration of Response (DOR)
Description: DOR is from first response (complete response (CR), CR unconfirmed (CRu) or partial response (PR)) to progression (PD) or death. Those without PD or death were censored at the last assessment.
  CR via PET-CT: Lymph/extralymph: Score 1/2/3a w/w-out resid mass, no new lesions, No FDG-avid disease in bone marrow (BM) CR via CT scan: Lymph/extralymph: Target/nodal ≤ 1.5 cm, no new lesions, normal BM CR Cohort 5: No contrast enhance, no corticosteroid, normal eye exam, neg CSF cytology CRu Cohort 5: No contrast enhance, min abnorm, normal eye exam, neg CSF cytology PR via PET-CT: Lymph/extralymph: Score 4/5b, red uptake, no new lesions, resid uptake incr, reduced in BM PR via CT scan: Lymph/extralymph: 50% decr in sum of diam ≤ 6 target/extranodal, no new/nonmeasured lesions, Organ enlarge: Spleen decr > 50% PR Cohort 5: 50% decr in enhancing tumor, no contrast enhance, Eye exam: Minor abnorm, decr in vitreous cells/retinal infiltrate, negative, persist or suspic CSF cytology.
Time Frame: From JCAR017 infusion until disease progression, death due to any reason, end of study, the start of another anticancer therapy, or hemopoietic stem cell transplant (HSCT) (up to approximately 63 months)
Population: All participants in the JCAR017 treated set who achieved a best overall response of complete response (and/ or CRu in cohort 5) or partial response/ remission.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 24 | 20 | 7 | 1 | 4 | 8
Months | 3.83 [2.07 to 17.05] | 3.91 [1.87 to NA] — Insufficient number of events to calculate upper limit of the CI using the K-M method. | 9.07 [2.04 to NA] — Insufficient number of events to calculate upper limit of the CI using the K-M method. | 17.97 [17.97 to 17.97] | 17.63 [2.46 to 23.10] | NA [2.69 to NA] — Insufficient number of events to calculate median and upper limit of the CI using the K-M method.

18. Secondary Outcome: Maximum Concentration (Cmax) of JCAR017 by qPCR
Description: Cmax is the maximum or peak concentration of drug reached in the plasma following a dose of the drug.
  Quantitative polymerase chain reaction (qPCR) was used to determine Cmax by detecting the JCAR017 transgene.
  Baseline is defined as the last available recorded value on or prior to the date of JCAR017 infusion.
Time Frame: At baseline and up until 24 months post JCAR017 infusion
Population: All participants in the JCAR017 treated set with baseline and on-study PK measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies/ug
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 34 | 22 | 10 | 1 | 5 | 9
Copies/ug | 23132.1 (434.6) | 21960.0 (278.1) | 17337.8 (894.4) | 51121.0 (NA) — Insufficient number of participants to calculate Geometric Coefficient of Variation. | 7661.6 (1730.0) | 32027.1 (101.4)

19. Secondary Outcome: Time to Peak Concentration (Tmax) of JCAR017 by qPCR
Description: Time to maximum concentration (Tmax) is the time it takes for a drug to reach the maximum concentration (Cmax) after administration.
  Quantitative polymerase chain reaction (qPCR) was used to determine Tmax by detecting the JCAR017 transgene.
  Baseline is defined as the last available recorded value on or prior to the date of JCAR017 infusion.
Time Frame: At baseline and up until 24 months post JCAR017 infusion
Population: All participants in the JCAR017 treated set with baseline and on-study PK measurements.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 34 | 22 | 10 | 1 | 5 | 9
Days | 11.6 [3.0 to 28.0] | 9.0 [7.0 to 14.0] | 84.1 [7.0 to 733.0] | 10.0 [10.0 to 10.0] | 9.0 [7.0 to 14.0] | 12.2 [10.0 to 21.0]

20. Secondary Outcome: Total Exposure to JCAR017 as Measured by Area Under the Curve (AUC) of JCAR017 by qPCR
Description: Area Under the Curve (AUC) represents the total exposure of participants to study drug.
  Quantitative polymerase chain reaction (qPCR) was used to determine AUC by detecting the JCAR017 transgene.
  Baseline is defined as the last available recorded value on or prior to the date of JCAR017 infusion.
Time Frame: At baseline and up until 24 months post JCAR017 infusion
Population: All participants in the JCAR017 treated set with baseline and on-study PK measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*copies/ug
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 34 | 22 | 10 | 1 | 5 | 9
Days*copies/ug | 185586.667 (325.6) | 157499.362 (211.9) | 134819.085 (1268.9) | 286119.439 (NA) — Insufficient number of participants to calculate Geometric Coefficient of Variation. | 64945.715 (1345.7) | 199731.737 (136.8)

21. Secondary Outcome: Percent of Participants With Presence of JCAR017 Transgene in Peripheral Blood by qPCR
Description: Persistence is defined as a transgene count greater than or equal to the lower limit of detection (LLOD) of 5 copies per reaction. Data obtained after the start of a new anti-cancer therapy were excluded. qPCR = Quantitative polymerase chain reaction.
Time Frame: At Day 29 and Months 2, 3, 6, 9, 12, 18, and 24 post JCAR017 infusion.
Population: All participants in the JCAR017 treated set with baseline and on-study JCAR017 transgene results.
Measure: Number; unit: Percent of Participants
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 34 | 21 | 10 | 1 | 5 | 9
Percent of Participants
  Day 29 | 88.2 | 95.2 | 100.0 | 100.0 | 80.0 | 100.0
  Month 2: number analyzed (Participants) | 30 | 18 | 7 | 1 | 4 | 8
  Month 2 | 70.0 | 66.7 | 100.0 | 100.0 | 100.0 | 62.5
  Month 3: number analyzed (Participants) | 26 | 16 | 7 | 1 | 4 | 8
  Month 3 | 61.5 | 50.0 | 100.0 | 100.0 | 100.0 | 37.5
  Month 6: number analyzed (Participants) | 12 | 11 | 7 | 1 | 3 | 6
  Month 6 | 33.3 | 45.5 | 71.4 | 0.0 | 100.0 | 16.7
  Month 9: number analyzed (Participants) | 12 | 5 | 5 | 1 | 3 | 4
  Month 9 | 41.7 | 40.0 | 60.0 | 0.0 | 100.0 | 25.0
  Month 12: number analyzed (Participants) | 10 | 7 | 4 | 1 | 3 | 4
  Month 12 | 40.0 | 57.1 | 100.0 | 0.0 | 66.7 | 0.0
  Month 18: number analyzed (Participants) | 8 | 7 | 4 | 1 | 2 | 5
  Month 18 | 25.0 | 57.1 | 75.0 | 0.0 | 100.0 | 20.0
  Month 24: number analyzed (Participants) | 7 | 6 | 3 | 1 | 2 | 5
  Month 24 | 28.6 | 50.0 | 100.0 | 0.0 | 100.0 | 20.0

22. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer - Quality of Life C30 Questionnaire (EORTC QLQ-C30) Scores
Description: The EORTC QLQ-C30 consists of five functional scales (physical, role, emotional, cognitive, social), three symptom scales (fatigue, nausea/vomiting, pain), a global health status/health-related quality of life (HRQoL) scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties). The questionnaire is scored on a 4-point Likert scale: 1 = not at all, 2 = a little, 3 = quite a bit, 4 = very much. The raw score is the average of the items contributing to the scale. The final scores are calculated via linear transformation of raw scores and range from 0 to 100. For functional scales higher scores indicate better QoL. For symptom scales and single items lower scores indicate fewer symptoms, i.e. better QoL. Baseline the last available recorded scores on or prior to the date of JCAR017 infusion. Only global health, fatigue, physical and cognitive functioning subscales were assessed.
Time Frame: At baseline and Day 1, 29, 60, 90, 180, 270, 365, 545, and 730 post JCAR017 infusion.
Population: All participants in the JCAR017-treated set with completed baseline questionnaires and with at least one completed post-baseline questionnaire.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 34 | 23 | 10 | 1 | 5 | 9
Scores on a Scale
  Global Health Status: Change from baseline Day 1 | -4.41 (17.070) | -5.07 (17.898) | -6.67 (10.244) | -8.33 (NA) — Insufficient number of participants to calculate standard deviation. | 8.33 (25.685) | -7.41 (12.108)
  Global Health Status: Change from baseline Day 29: number analyzed (Participants) | 33 | 19 | 10 | 1 | 4 | 9
  Global Health Status: Change from baseline Day 29 | -1.26 (14.301) | 0.00 (18.002) | -4.17 (17.236) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 16.67 (11.785) | -1.85 (14.299)
  Global Health Status: Change from baseline Day 60: number analyzed (Participants) | 30 | 17 | 6 | 1 | 3 | 9
  Global Health Status: Change from baseline Day 60 | 5.00 (14.778) | 7.84 (17.547) | 4.17 (16.457) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 13.89 (26.788) | 9.26 (8.784)
  Global Health Status: Change from baseline Day 90: number analyzed (Participants) | 27 | 13 | 7 | 1 | 3 | 9
  Global Health Status: Change from baseline Day 90 | 2.47 (14.766) | 1.28 (22.527) | -5.95 (17.817) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 22.22 (41.107) | 4.63 (8.448)
  Global Health Status: Change from baseline Day 180: number analyzed (Participants) | 12 | 8 | 7 | 1 | 3 | 6
  Global Health Status: Change from baseline Day 180 | 6.94 (13.685) | 1.04 (23.332) | -13.10 (35.635) | -16.67 (NA) — Insufficient number of participants to calculate standard deviation. | 25.00 (22.048) | 2.78 (8.607)
  Global Health Status: Change from baseline Day 270: number analyzed (Participants) | 12 | 6 | 5 | 1 | 3 | 5
  Global Health Status: Change from baseline Day 270 | 6.25 (20.140) | 9.72 (9.742) | -3.33 (26.745) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 25.00 (22.048) | 3.33 (9.501)
  Global Health Status: Change from baseline Day 365: number analyzed (Participants) | 10 | 7 | 4 | 1 | 3 | 5
  Global Health Status: Change from baseline Day 365 | -6.67 (20.337) | 3.57 (11.664) | -12.50 (25.909) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 30.56 (26.788) | 3.33 (7.454)
  Global Health Status: Change from baseline Day 545: number analyzed (Participants) | 9 | 7 | 3 | 1 | 2 | 5
  Global Health Status: Change from baseline Day 545 | -6.48 (18.530) | 3.57 (26.726) | -5.56 (24.056) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 0.00 (47.140) | 1.67 (9.129)
  Global Health Status: Change from baseline Day 730: number analyzed (Participants) | 12 | 6 | 4 | 1 | 2 | 4
  Global Health Status: Change from baseline Day 730 | -11.11 (12.975) | -4.17 (12.638) | -6.25 (7.979) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 20.83 (29.463) | -2.08 (21.916)
  Physical Functioning: Change from baseline Day 1 | -3.33 (20.970) | -6.09 (21.074) | -3.33 (11.440) | -6.67 (NA) — Insufficient number of participants to calculate standard deviation. | -2.67 (19.777) | -3.70 (14.948)
  Physical Functioning: Change from baseline Day 29: number analyzed (Participants) | 33 | 19 | 10 | 1 | 5 | 9
  Physical Functioning: Change from baseline Day 29 | -2.63 (18.555) | -4.21 (10.706) | -10.00 (14.824) | 6.67 (NA) — Insufficient number of participants to calculate standard deviation. | -8.33 (16.667) | -8.15 (18.493)
  Physical Functioning: Change from baseline Day 60: number analyzed (Participants) | 30 | 17 | 6 | 1 | 3 | 9
  Physical Functioning: Change from baseline Day 60 | 3.11 (15.135) | -0.39 (21.275) | -4.44 (15.587) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | -2.22 (10.184) | -2.96 (10.062)
  Physical Functioning: Change from baseline Day 90: number analyzed (Participants) | 27 | 13 | 7 | 1 | 3 | 9
  Physical Functioning: Change from baseline Day 90 | 3.46 (16.781) | 3.59 (12.054) | -5.71 (11.174) | 6.67 (NA) — Insufficient number of participants to calculate standard deviation. | 11.11 (23.413) | -0.74 (18.692)
  Physical Functioning: Change from baseline Day 180: number analyzed (Participants) | 12 | 8 | 7 | 1 | 3 | 6
  Physical Functioning: Change from baseline Day 180 | 7.78 (12.975) | -8.33 (31.219) | -5.71 (19.024) | -6.67 (NA) — Insufficient number of participants to calculate standard deviation. | 15.56 (27.756) | -2.22 (24.825)
  Physical Functioning: Change from baseline Day 270: number analyzed (Participants) | 12 | 6 | 5 | 1 | 3 | 5
  Physical Functioning: Change from baseline Day 270 | 3.33 (10.050) | 1.11 (19.052) | -2.67 (22.410) | 6.67 (NA) — Insufficient number of participants to calculate standard deviation. | 24.44 (27.756) | -6.67 (31.972)
  Physical Functioning: Change from baseline Day 365: number analyzed (Participants) | 10 | 7 | 4 | 1 | 3 | 5
  Physical Functioning: Change from baseline Day 365 | 0.67 (16.163) | 0.95 (16.069) | -16.67 (20.000) | 6.67 (NA) — Insufficient number of participants to calculate standard deviation. | 22.22 (26.943) | 5.33 (11.926)
  Physical Functioning: Change from baseline Day 545: number analyzed (Participants) | 9 | 7 | 3 | 1 | 2 | 5
  Physical Functioning: Change from baseline Day 545 | -3.70 (26.690) | -1.90 (19.135) | -13.33 (23.094) | 6.67 (NA) — Insufficient number of participants to calculate standard deviation. | 13.33 (47.140) | 9.33 (11.155)
  Physical Functioning: Change from baseline Day 730: number analyzed (Participants) | 12 | 6 | 4 | 1 | 2 | 4
  Physical Functioning: Change from baseline Day 730 | 1.11 (15.785) | -8.89 (28.493) | -3.33 (8.607) | 6.67 (NA) — Insufficient number of participants to calculate standard deviation. | 3.33 (42.426) | -3.33 (11.547)
  Cognitive Functioning: Change from baseline Day 1 | -3.43 (17.301) | -3.62 (17.376) | -1.67 (9.461) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | -3.33 (13.944) | -1.85 (10.015)
  Cognitive Functioning: Change from baseline Day 29: number analyzed (Participants) | 33 | 19 | 10 | 1 | 4 | 9
  Cognitive Functioning: Change from baseline Day 29 | -2.53 (16.203) | 3.51 (14.250) | 3.33 (13.147) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 8.33 (21.517) | -7.41 (12.108)
  Cognitive Functioning: Change from baseline Day 60: number analyzed (Participants) | 30 | 17 | 6 | 1 | 3 | 9
  Cognitive Functioning: Change from baseline Day 60 | 2.78 (12.444) | 0.98 (10.978) | 0.00 (27.889) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 33.33 (44.096) | -1.85 (13.029)
  Cognitive Functioning: Change from baseline Day 90: number analyzed (Participants) | 27 | 13 | 7 | 1 | 3 | 9
  Cognitive Functioning: Change from baseline Day 90 | 0.00 (13.074) | -1.28 (12.659) | 4.76 (20.893) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 11.11 (19.245) | 0.00 (8.333)
  Cognitive Functioning: Change from baseline Day 180: number analyzed (Participants) | 12 | 8 | 7 | 1 | 3 | 6
  Cognitive Functioning: Change from baseline Day 180 | -2.78 (15.624) | -2.08 (5.893) | 11.90 (20.893) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 16.67 (28.868) | -5.56 (8.607)
  Cognitive Functioning: Change from baseline Day 270: number analyzed (Participants) | 12 | 6 | 5 | 1 | 3 | 5
  Cognitive Functioning: Change from baseline Day 270 | 0.00 (22.473) | 0.00 (0.000) | 3.33 (13.944) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 33.33 (44.096) | 3.33 (7.454)
  Cognitive Functioning: Change from baseline Day 365: number analyzed (Participants) | 10 | 7 | 4 | 1 | 3 | 5
  Cognitive Functioning: Change from baseline Day 365 | -11.67 (22.292) | 0.00 (0.000) | -4.17 (8.333) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | 22.22 (38.490) | 6.67 (9.129)
  Cognitive Functioning: Change from baseline Day 545: number analyzed (Participants) | 9 | 7 | 3 | 1 | 2 | 5
  Cognitive Functioning: Change from baseline Day 545 | -7.41 (18.840) | 2.38 (11.501) | -5.56 (19.245) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | -41.67 (82.496) | 3.33 (7.454)
  Cognitive Functioning: Change from baseline Day 730: number analyzed (Participants) | 12 | 6 | 4 | 1 | 2 | 4
  Cognitive Functioning: Change from baseline Day 730 | -1.39 (18.060) | -5.56 (8.607) | -4.17 (15.957) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | -16.67 (23.570) | -4.17 (8.333)
  Fatigue: Change from baseline Day 1 | 1.63 (26.959) | 1.45 (16.173) | 3.33 (20.320) | 0.00 (NA) — Insufficient number of participants to calculate standard deviation. | -20.00 (30.832) | 1.23 (18.794)
  Fatigue: Change from baseline Day 29: number analyzed (Participants) | 33 | 19 | 10 | 1 | 4 | 9
  Fatigue: Change from baseline Day 29 | 3.03 (24.418) | 2.34 (12.046) | 5.56 (17.568) | -11.11 (NA) — Insufficient number of participants to calculate standard deviation. | -13.89 (27.778) | 6.17 (14.815)
  Fatigue: Change from baseline Day 60: number analyzed (Participants) | 30 | 17 | 6 | 1 | 3 | 9
  Fatigue: Change from baseline Day 60 | -9.63 (18.623) | -1.31 (20.743) | 3.70 (31.946) | 11.11 (NA) — Insufficient number of participants to calculate standard deviation. | -14.81 (35.717) | 0.00 (17.568)
  Fatigue: Change from baseline Day 90: number analyzed (Participants) | 27 | 13 | 7 | 1 | 3 | 9
  Fatigue: Change from baseline Day 90 | -4.53 (19.795) | -4.27 (17.881) | 4.76 (35.635) | -11.11 (NA) — Insufficient number of participants to calculate standard deviation. | -37.04 (12.830) | -3.70 (22.906)
  Fatigue: Change from baseline Day 180: number analyzed (Participants) | 12 | 8 | 7 | 1 | 3 | 6
  Fatigue: Change from baseline Day 180 | -8.33 (21.254) | 2.78 (34.503) | -4.76 (38.946) | 22.22 (NA) — Insufficient number of participants to calculate standard deviation. | -37.04 (23.130) | 0.00 (33.702)
  Fatigue: Change from baseline Day 270: number analyzed (Participants) | 12 | 6 | 5 | 1 | 3 | 5
  Fatigue: Change from baseline Day 270 | -9.26 (15.594) | 0.00 (22.222) | -6.67 (14.907) | -11.11 (NA) — Insufficient number of participants to calculate standard deviation. | -29.63 (42.066) | -2.22 (34.605)
  Fatigue: Change from baseline Day 365: number analyzed (Participants) | 10 | 7 | 4 | 1 | 3 | 5
  Fatigue: Change from baseline Day 365 | -3.33 (14.861) | -4.76 (20.141) | 13.89 (33.179) | -11.11 (NA) — Insufficient number of participants to calculate standard deviation. | -44.44 (22.222) | -13.33 (14.487)
  Fatigue: Change from baseline Day 545: number analyzed (Participants) | 9 | 7 | 3 | 1 | 2 | 5
  Fatigue: Change from baseline Day 545 | 4.94 (25.526) | -1.59 (19.698) | -3.70 (27.962) | -11.11 (NA) — Insufficient number of participants to calculate standard deviation. | -5.56 (23.570) | -11.11 (15.713)
  Fatigue: Change from baseline Day 730: number analyzed (Participants) | 12 | 6 | 4 | 1 | 2 | 4
  Fatigue: Change from baseline Day 730 | 0.93 (22.947) | 3.70 (9.072) | 5.56 (14.344) | -11.11 (NA) — Insufficient number of participants to calculate standard deviation. | -16.67 (7.857) | -8.33 (16.667)

23. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Treatment-Lymphoma "Additional Concerns" Subscale (FACT-LymS) Scores
Description: The Functional Assessment of Cancer Treatment-Lymphoma "Additional concerns" subscale (FACT-LymS) consists of the FACT-General scale and a 15-item lymphoma-specific additional concerns subscale (LYM). This scale addresses symptoms and functional limitations that are important to lymphoma patients. Only the LYM subscale was administered in this study. The LYM items are scored on a 0 ("Not at all") to 4 ("Very much") response scale. Items are aggregated to a single score on a 0-60 scale. Lower scores indicate better health outcomes. Baseline the last available recorded scores on or prior to the date of JCAR017 infusion.
Time Frame: At baseline and Day 1, 29, 60, 90, 180, 270, 365, 545, and 730 post JCAR017 infusion.
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
Number analyzed (Participants) | 33 | 23 | 10 | 1 | 5 | 9
Scores on a Scale
  Change from baseline Day 1 | 0.7 (8.17) | 0.1 (7.05) | 1.9 (5.92) | 1.0 (NA) — Insufficient number of participants to calculate standard deviation. | -4.0 (6.52) | -1.2 (11.08)
  Change from baseline Day 29: number analyzed (Participants) | 33 | 19 | 10 | 1 | 4 | 9
  Change from baseline Day 29 | -1.7 (7.14) | -2.7 (4.56) | 1.3 (7.24) | -4.0 (NA) — Insufficient number of participants to calculate standard deviation. | -6.5 (8.10) | 1.0 (9.08)
  Change from baseline Day 60: number analyzed (Participants) | 30 | 17 | 6 | 1 | 3 | 9
  Change from baseline Day 60 | -2.8 (5.42) | -2.0 (4.20) | -3.3 (9.99) | -4.0 (NA) — Insufficient number of participants to calculate standard deviation. | -4.7 (8.33) | -0.4 (9.95)
  Change from baseline Day 90: number analyzed (Participants) | 27 | 13 | 7 | 1 | 3 | 9
  Change from baseline Day 90 | -0.4 (5.42) | -2.8 (3.83) | 0.6 (9.25) | -5.0 (NA) — Insufficient number of participants to calculate standard deviation. | -6.7 (8.50) | -1.7 (8.67)
  Change from baseline Day 180: number analyzed (Participants) | 12 | 8 | 7 | 1 | 3 | 6
  Change from baseline Day 180 | 0.6 (5.14) | -1.8 (5.65) | -3.6 (10.20) | 2.0 (NA) — Insufficient number of participants to calculate standard deviation. | -8.0 (7.00) | 1.0 (7.27)
  Change from baseline Day 270: number analyzed (Participants) | 12 | 6 | 5 | 1 | 3 | 5
  Change from baseline Day 270 | -0.3 (6.78) | -3.7 (2.25) | -1.0 (10.07) | -8.0 (NA) — Insufficient number of participants to calculate standard deviation. | -10.00 (12.53) | 2.4 (5.22)
  Change from baseline Day 365: number analyzed (Participants) | 10 | 7 | 4 | 1 | 3 | 5
  Change from baseline Day 365 | 1.3 (7.01) | -3.3 (3.30) | 2.0 (12.03) | -6.0 (NA) — Insufficient number of participants to calculate standard deviation. | -6.7 (10.69) | 1.4 (7.33)
  Change from baseline Day 545: number analyzed (Participants) | 9 | 7 | 3 | 1 | 2 | 5
  Change from baseline Day 545 | 0.7 (7.14) | -3.7 (4.35) | -4.7 (4.16) | -3.0 (NA) — Insufficient number of participants to calculate standard deviation. | 3.5 (6.36) | -1.0 (4.85)
  Change from baseline Day 730: number analyzed (Participants) | 12 | 6 | 4 | 1 | 2 | 4
  Change from baseline Day 730 | 1.4 (7.12) | -0.8 (1.33) | -1.8 (5.32) | -2.0 (NA) — Insufficient number of participants to calculate standard deviation. | -1.5 (12.02) | -1.5 (1.29)

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events from their date of leukapheresis until their study completion (assessed up to approximately 63 months).
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that underwent leukapheresis and may or may not have received at least 1 dose of JCAR017.
Arm/Group | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma | Cohort 5: Primary Central Nervous System Lymphoma | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting
All-Cause Mortality (participants affected / at risk) | 32/45 | 22/32 | 9/14 | 0/4 | 5/7 | 4/11
Serious Adverse Events (participants affected / at risk) | 19/45 | 8/32 | 2/14 | 0/4 | 2/7 | 1/11
Other Adverse Events (participants affected / at risk) | 40/45 | 25/32 | 12/14 | 1/4 | 5/7 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy (N=45) | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy (N=32) | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 (N=14) | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma (N=4) | Cohort 5: Primary Central Nervous System Lymphoma (N=7) | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 7 | 1 | 0 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Candida sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 4 | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 0 | 0 | 1 | 0
Stupor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 5 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 5 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Diffuse B-cell Lymphoma Who Failed ≥ 2 Lines of Therapy (N=45) | Cohort 2: Transplant Ineligible Diffuse B-cell Lymphoma Who Failed First Line Therapy (N=32) | Cohort 3: Japan Specific - Meeting Eligibility Criteria for Cohort 1 or 2 (N=14) | Cohort 4: Newly Diagnosed High-Grade B-cell Lymphoma (N=4) | Cohort 5: Primary Central Nervous System Lymphoma (N=7) | Cohort 7: Meeting Cohort 1 Criteria Suitable for Treatment in an Outpatient Setting (N=11)
Acquired antithrombin III deficiency (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 21 | 8 | 10 | 0 | 3 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 1 | 0 | 0 | 0 | 0
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 | 0 | 4 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 9 | 5 | 11 | 0 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 9 | 4 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 35 | 22 | 11 | 1 | 5 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 11 | 11 | 1 | 3 | 3
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Keratopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 7 | 2 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 2 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 6 | 3 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 3 | 2 | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 4 | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 5 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 20 | 10 | 2 | 0 | 2 | 1
Cytokine release syndrome (Immune system disorders) | 12 | 12 | 6 | 0 | 3 | 0
Hypogammaglobulinaemia (Immune system disorders) | 6 | 3 | 4 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 3 | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 1 | 1 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 1 | 0
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 7 | 4 | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT03484702/Prot_SAP_000.pdf